CLINICAL TRIAL: NCT01581931
Title: Bioequivalence of Metformin Under Fed Conditions After Administration of a 2.5 mg Linagliptin / 500 mg Metformin Fixed Dose Combination Tablet Compared With Single Linagliptin 2.5 mg and Metformin 500 mg Tablets Administered Together in Healthy Male and Female Volunteers, (an Open-label, Randomised, Single Dose, Two-way Crossover, Phase I Trial)
Brief Title: Bioequivalence of Metformin Under Fed Conditions After Administration of Linagliptin / Metformin Fixed Dose Combination Tablet and Single Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.20; 2011-005423-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Results first posted 2013-08-20 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Metformin

ARMS (2):
- Linagliptin/metformin (Experimental): fixed dose combination tablet (FDC)
  Interventions: Drug: Linagliptin/metformin
- Linagliptin and metformin (Experimental): single tablets
  Interventions: Drug: Metformin; Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin/metformin — FDC
  Arms: Linagliptin/metformin
Drug: Metformin — single tablet Metformin
  Arms: Linagliptin and metformin
Drug: Linagliptin — single tablet Linagliptin
  Arms: Linagliptin and metformin

SUMMARY:
To establish bioequivalence (BE) under fed conditions between metformin in linagliptin/metformin fixed dose combination tablet and metformin reference product administered in free combination togther with linagliptin

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1288.20.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Lina+Met Single Tablets / Lina+Met FDC Tablet: Subjects are treated with single linagliptin 2.5 mg and metformin 500 mg tablets in the first period. After a washout period of at least 35 days, the subjects are treated with a 2.5 mg linagliptin / 500 mg metformin fixed-dose-combination (FDC) tablet in period 2.
- Lina+Met FDC Tablet / Lina+Met Single Tablets: Subjects are treated with a 2.5 mg linagliptin / 500 mg metformin fixed-dose-combination (FDC) tablet in the first period. After a washout period of at least 35 days, the subjects are treated with single linagliptin 2.5 mg and metformin 500 mg tablets in period 2.
Period: First Period
Arm/Group | Lina+Met Single Tablets / Lina+Met FDC Tablet | Lina+Met FDC Tablet / Lina+Met Single Tablets
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout
Arm/Group | Lina+Met Single Tablets / Lina+Met FDC Tablet | Lina+Met FDC Tablet / Lina+Met Single Tablets
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Period
Arm/Group | Lina+Met Single Tablets / Lina+Met FDC Tablet | Lina+Met FDC Tablet / Lina+Met Single Tablets
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This was an open-label, randomised, single dose, 2-way crossover trial with 2 treatments and 2 treatment sequences. The single dose administrations in each treatment period were separated by a washout period of at least 35 days.
Arm/Group | Overall Study
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 38.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 15

OUTCOME MEASURES:

1. Secondary Outcome: Area Under Curve From 0 to Infinity Hours (AUC0-infty) of Metformin
Description: AUC0-infty represents the area under the concentration curve of metformin in plasma from time 0 extrapolated to infinity. Note, the geometric mean is actually an adjusted geometric mean.
Time Frame: 0:20, 0:40, 1, 1:30, 2, 3, 4, 5, 6, 8, 12, 24, 34, 48, 72 hours
Population: Treated set - all subjects taking at least 1 dose of trial medication
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Groups:
- Lina+Met Single Tablets: Subjects are treated with single linagliptin 2.5 mg and metformin 500 mg tablets
- Lina+Met FDC Tablet: Subjects are treated with a 2.5 mg linagliptin / 500 mg metformin fixed-dose-combination (FDC) tablet
Arm/Group | Lina+Met Single Tablets | Lina+Met FDC Tablet
Number analyzed (Participants) | 30 | 32
ng·h/mL | 7343.59 (9.7) | 7174.30 (9.7)
Statistical Analysis 1: Comparison: Lina+Met Single Tablets vs Lina+Met FDC Tablet; Test type: Non-Inferiority or Equivalence — Equivalence margin: the 90% confidence intervall has to be within the intervall (80%, 125%); ANOVA; Adjusted geometric mean ratio = 97.69, 95% CI 2-sided [93.63 to 101.94], Standard Deviation 9.7 — Numerator: FDC tablet; denominator: single tablets of linagliptin and metformin; The dispersion parameter is actually the geometric coefficient of variation

2. Secondary Outcome: Time to Maximum Concentration (Tmax) of Metformin
Description: Time from dosing to the maximum concentration of metformin in plasma.
Time Frame: 0:20, 0:40, 1, 1:30, 2, 3, 4, 5, 6, 8, 12, 24, 34, 48, 72 hours
Population: Treated set - all subjects taking at least 1 dose of trial medication
Measure: Median (Full Range); unit: Hours
Arm/Group | Lina+Met Single Tablets | Lina+Met FDC Tablet
Number analyzed (Participants) | 30 | 32
Hours | 4.00 [2.00 to 6.00] | 4.00 [1.00 to 6.00]

3. Secondary Outcome: Terminal Half-life t1/2 of Metformin
Description: The terminal half-life of metformin in plasma is denoted by t1/2.
Time Frame: 0:20, 0:40, 1, 1:30, 2, 3, 4, 5, 6, 8, 12, 24, 34, 48, 72 hours
Population: Treated set - all subjects taking at least 1 dose of trial medication
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Lina+Met Single Tablets | Lina+Met FDC Tablet
Number analyzed (Participants) | 30 | 32
Hours | 9.14 (87.4) | 8.03 (86.0)

4. Primary Outcome: Area Under Curve From 0 to tz Hours (AUC0-tz) of Metformin
Description: AUC0-tz represents the area under the concentration curve of metformin in plasma from 0 to the time of the last quantifiable plasma contentration of the analyte. Note, the geometric mean is actually an adjusted geometric mean.
Time Frame: 0:20, 0:40, 1, 1:30, 2, 3, 4, 5, 6, 8, 12, 24, 34, 48, 72 hours
Population: Treated set - all subjects taking at least 1 dose of trial medication
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | Lina+Met Single Tablets | Lina+Met FDC Tablet
Number analyzed (Participants) | 30 | 32
ng·h/mL | 7219.03 (9.8) | 7057.52 (9.8)
Statistical Analysis 1: Comparison: Lina+Met Single Tablets vs Lina+Met FDC Tablet; Test type: Non-Inferiority or Equivalence — Equivalence margin: the 90% confidence intervall has to be within the intervall (80%, 125%); ANOVA; Adjusted geometric mean ratio = 97.76, 90% CI 2-sided [93.64 to 102.07], Standard Deviation 9.8 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Maximum Concentration (Cmax) of Metformin
Description: Cmax represents the maximum concentration of metformin in plasma. Note, the geometric mean is actually an adjusted geometric mean.
Time Frame: 0:20, 0:40, 1, 1:30, 2, 3, 4, 5, 6, 8, 12, 24, 34, 48, 72 hours
Population: Treated set - all subjects taking at least 1 dose of trial medication
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lina+Met Single Tablets | Lina+Met FDC Tablet
Number analyzed (Participants) | 30 | 32
ng/mL | 855.09 (10.0) | 844.72 (10.0)
Statistical Analysis 1: Comparison: Lina+Met Single Tablets vs Lina+Met FDC Tablet; Test type: Non-Inferiority or Equivalence — Equivalence margin: the 90% confidence intervall has to be within the intervall (80%, 125%); ANOVA; Adjusted geometric mean ratio = 98.79, 90% CI 2-sided [94.55 to 103.21], Standard Deviation 10.0 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: First treatment with study drug until End-of-Study (which was within 4 to 14 days after last study drug administration), i.e., 39 to 49 days after first treatment with study drug.
Arm/Group | Lina+Met Single Tablets | Lina+Met FDC Tablet
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/32
Other Adverse Events (participants affected / at risk) | 6/31 | 9/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lina+Met Single Tablets (N=31) | Lina+Met FDC Tablet (N=32)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lina+Met Single Tablets (N=31) | Lina+Met FDC Tablet (N=32)
Nasopharyngitis (Infections and infestations) | 0 | 2
Headache (Nervous system disorders) | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.